CLINICAL TRIAL: NCT00206011
Title: Open Versus Endoscopic Surgery of Condylar Neck Fractures
Brief Title: Open Versus Endoscopic Surgery of Craniomaxillofacial (CMF) Condylar Neck Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-CMF-01
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Condylar Neck Fractures
Keywords: Condylar neck; fractures; endoscopic; Helkimo Dysfunction index
MeSH Terms: conditions — Fractures, Bone | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: Endoscopic surgery
- 2 (Other)
  Interventions: Procedure: Endoscopic surgery

INTERVENTIONS:
Procedure: Endoscopic surgery — Open surgical intervention compared to endoscopic intervention

SUMMARY:
This study is a comparison of open surgery versus an endoscopic approach in condylar neck fractures; it will look at functional outcome, cosmetic outcome and patient satisfaction.

DETAILED DESCRIPTION:
The primary outcome measure is functional outcome based on the Helkimo dysfunction index.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient > 18 years
* Unilateral or bilateral fracture of the condylar neck
* Inclination of the condyle > 30%
* Severe dislocation
* Severe pain upon palpation/movement
* Eligible for open reduction and internal fixation of the fracture
* Amenable to endoscopic as well as open surgery

Exclusion Criteria:

* High or intracapsular condylar neck fracture
* Very low fractures that can be reduced intraorally
* CMF malfunctioning
* Drug or alcohol abuse
* General or local conditions that adversely affect bone physiology
* Physical or mental incapacity to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2003-04; Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Functional outcome based on the Helkimo dysfunction index | 3 months

SECONDARY OUTCOMES:
Complication rate | 24 months
Cost effectiveness | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Schmlezeisen, Prof. Dr., Principal Investigator — Universitaet Freiburg
Locations (1):
- Universitaestklinik Freiburg, Klinik für Mund- Gesichts- und Kieferchirurgie, Freiburg im Breisgau, Germany